CLINICAL TRIAL: NCT06414109
Title: Mindfulness-Based Intervention for Adolescents With Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-2359
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Migraine; Migraine in Adolescence
Keywords: Adolescent; Mindfulness; Mindfulness Intervention; Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BREATHE-Migraine (Experimental): Participants will receive 6 weekly 1-hour sessions of a remotely-delivered mindfulness-based intervention in a group setting.
  Interventions: Behavioral: BREATHE-Migraine

INTERVENTIONS:
Behavioral: BREATHE-Migraine — The BREATHE-Migraine intervention was adapted from the research-supported curriculum, "Learning to BREATHE" (Broderick, 2021), based on qualitative feedback from adolescents with migraine, their parents, and pediatric headache providers. BREATHE-Migraine includes experiential and didactic exercises designed to address emotion regulation and the stress of living with frequent migraine.

SUMMARY:
The goal of this study is to assess feasibility and acceptability of a mindfulness-based intervention adapted for adolescents with migraine to inform a future randomized trial assessing effects of the intervention on headache-related outcomes.

DETAILED DESCRIPTION:
Mindfulness-based intervention (MBI) shows promise in adults with migraine, but research is limited in adolescents. The current study aims to advance behavioral treatments for adolescents with frequent migraine by adapting an existing empirically-supported MBI for adolescents (Learning to BREATHE) to meet the unique needs of adolescents with chronic migraine. In Phase I of the study, we will use feedback solicited from interviews with teens with chronic migraine, their parents, and healthcare providers documenting the experience of living with chronic migraine and on the content and delivery of the MBI to create an adapted telehealth group intervention specifically tailored for adolescents with frequent migraine. In Phase II of the study, the adapted MBI will be piloted in a single-arm trial with adolescents with frequent migraine to assess feasibility, acceptability, and preliminary clinical signals.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 to 18 years
* Diagnosed with migraine by medical provider using criteria from the International Classification of Headache Disorders, Third Edition
* Patient report of >= 8 headache days per month
* PedMIDAS Score of > 10 (at least mild headache-related disability)

Exclusion Criteria:

* Major comorbid medical condition (e.g., cancer, epilepsy)
* Active psychosis or suicidal ideation
* Inability to provide consent/assent

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Intervention feasibility | Up to 6 weeks
  Percent of sessions attended; Qualitative data generated via focus group interviews (questions will include barriers and facilitators to completing the intervention)
Intervention acceptability | 7 weeks
  Ratings on program acceptability questionnaire (higher scores indicate higher acceptability); Qualitative data generated via focus group interviews (questions will include positive and negative perceptions of the intervention)

SECONDARY OUTCOMES:
Change in headache-related disability | Baseline, 6 weeks
  The Pediatric Migraine Disability Assessment (PedMIDAS) is a 6-item self-report questionnaire measuring the extent to which headaches interfered with school attendance and functioning, home functioning, and social attendance and functioning. Adolescents will be asked to indicate the number of days in the past 3 months in which they were unable to attend or fully participate in a range of activities. Lower scores indicate less disability.
Change in emotion regulation | Baseline, 6 weeks
  The Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) is an 18-item self-report measure of various dimensions of emotion dysregulation. Items are rated on a 6-point Likert scale ranging from 1 (almost never) to 5 (almost always). The DERS-SF provides a total score and 6 subscale scores. Lower scores indicate better emotion regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Clementi, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States